CLINICAL TRIAL: NCT03963245
Title: Project Meaningful Activities and Recovery (MA&R)
Brief Title: Project Meaningful Activities and Recovery
Acronym: MA&R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F-61171-15-05
Record Dates: First submitted 2019-04-16; First posted 2019-05-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Mental Illness
Keywords: Psychiatric Disabilities; Rehabilitation; Recovery; Occupational therapy; Peer-support
MeSH Terms: conditions — Mental Disorders | interventions — Salvage Therapy; Standard of Care; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): MA&R - an eight months rehabilitation intervention in addition to standard care and treatment in Community Mental Health Centres in Copenhagen, and psychiatric rehabilitation services in Copenhagen, Odense and Svendborg, Denmark
  Interventions: Behavioral: Meaningful Activities and Recovery; Behavioral: Standard Care and Treatment
- Control group (Active Comparator): Standard care and treatment in Community Mental Health Centres in Copenhagen, and psychiatric rehabilitation services in Copenhagen, Odense and Svendborg, Denmark
  Interventions: Behavioral: Standard Care and Treatment

INTERVENTIONS:
Behavioral: Meaningful Activities and Recovery — MA&R is a new rehabilitation program for people with psychiatric disabilities. MA&R aims to enable participation in everyday activities that are meaningful to the individual.
  MA&R is based on occupational science, and the underlying premise that there is a connection between mental health, recovery and meaningful everyday activities. The goal of MA&R is that participants through the course become better at connecting daily activities with values, interests, plans and goals. When this connection is strengthened, it supports the experience of meaningfulness in everyday life.
  MA&R is led by two mentors where one mentor is an occupational therapist (or similar) and the other has lived experiences of mental vulnerability and recovery.
  Arms: Intervention group
Behavioral: Standard Care and Treatment — For community mental health centres: medicine, psychoeducation, relational support, peer-support, psychotherapy, social counselling, care manager
  For psychiatric rehabilitation services in Copenhagen, Odense and Svendborg: drop in centres, relational support, skills training, peer-support

SUMMARY:
Occupational therapy interventions are often part of the treatment and rehabilitation services offered to people with mental illnesses. Occupational therapy can be an important contribution when the purpose is to promote participation in everyday activities that are meaningful for the individual. (1-3) There is limited evidence to support whether occupational therapy interventions for people with mental illnesses have an effect. (2,3) Based on principles from Lifestyle Redesign®, which is an evidence-based occupational therapy intervention for older people, a comparative qualitative study with participant experiences from various psychosocial rehabilitation efforts, and a dialogue-based collaboration with experienced occupational therapists and peer staff from community mental health centers, we developed a new recovery oriented occupational therapy intervention to people with disabilities due to mental illness.

The intervention "Meaningful activities and recovery" (MA&R) - is an eight-month rehabilitation program. The aim of MA&R is to enable participation in activities that are meaningful to the individual.

Project Meaningful Activities and Recovery (MA&R) is a clinical trial where the purpose is to compare the effects of: 1) "Meaningful activities and Recovery" (MA&R) in addition to standard care and 2) standard care as it is now offered to people with psychiatric disabilities.

The design is a randomized clinical trial with self-reported assessments. Based on sample size calculation, 128 participants will be included in the trials. The primary endpoint is activity engagement, and the secondary effect goals are personal recovery, functioning and quality of life. Participants are followed up at the end of the intervention, after eight months.

DETAILED DESCRIPTION:
Participants Participants are people, diagnosed with mental illness and who uses services in either community mental health centres in Copenhagen, or live in supported accommodations, or receive psychiatric rehabilitation services in Copenhagen, Odense or Svendborg, three Danish cities.

Recruitment The initial contact with the participants is done by staff at the community mental health centres, supported housings or rehabilitation services in Copenhagen, Odense and Svendborg, talking with relevant candidates based on the research project's inclusion and exclusion criteria and informing them orally and in writing about the research project. This is supplemented, with the approval of the sites, by hanging posters in common rooms and possibly. presentation by researcher to the resident group / patients / citizen group at joint meeting to encourage self-referral. People who are interested in participating in the research project (hereinafter referred to as potential participants) contact the researcher or notify this to staff who communicate contact with researcher on behalf of citizens. An appointment is made for information interviews and pre-screening. Potential participants are invited to bring relatives or a contact person to the appointment. The oral information is given before the written one, and it is ensured that the information conversation takes place undisturbed. The participant information is provided in the form of a folder with adequate information about the experiment. The potential participant is informed that participation in the trial is voluntary and should not have any side effects, and that at any time they may exit the trial, without consequence for future support and the right to psychiatric treatment or rehabilitation services.

If the prospective participant, after being informed of the research project, is still interested in participating in the research project, the researcher conducts a functional level assessment at Mini-ICF-APP and asks the potential participant whether he or she is diagnosed with a mental illness. Based on this, it is decided whether the potential participant can be included.

Then, a consent form is handed out. Three-day reflection time (at least 24 hours) is offered. The written consent will be dated and numbered with the participant number. The participant will receive a copy while the original will be archived in a locked cabinet and scanned electronically and stored on a logged drive.

When written consent is given, the researcher obtains data by asking the participant, ie. self-reporting socio-demographic data and information on the mental illness. The researcher sends questionnaires to the participant, either electronically or as a letter, depending on what the participant prefers.

All participants receive a serial number and data are entered in REDCap.

Randomization and blinding Participants who have given informed consent and who have completed the questionnaires (baseline data) are randomized to either the control group or the intervention group. Randomization is done in RedCap. It is randomized according to varying block sizes, unknown to the researcher. The researcher makes sure to inform the participant which group they have come in either directly or through referring staff.

The researcher, staff and participants are not blinded to which group the participant comes in. To ensure blindness in collecting follow-up data, these data are obtained by research assistants who are blinded on the allocation. Blinding of the researcher during the analysis phase and when drawing conclusions is ensured by the participants being provided with a new serial number before the analyzes begin and the intervention groups are indicated by a "x" and "y".

Interventions There are two types of interventions

1. MA&R in addition to standard services
2. Standard services

MA&R lasts eight months and consists of two courses, MA&R I and MA&R II, which are contemplated by each other. MA&R I supports a greater self-awareness of the importance of daily life activities and is primarily based on reflection and conversation. MA&R II is about anchoring new activities, habits or patterns of action in everyday life and is primarily action-oriented.

MA&R I consists of six group sessions and five individual meetings. The community sessions take place weekly and typically lasts two hours, with the possibility of shortening the meeting for one hour.

The MA&R II consists of five joint sessions and six dialogue meetings. As in MA&R I, the joint sessions and dialogue meetings take place alternately. For the joint sessions, the participants are presented with strategies and tools for enabling activity participation, for example, by promoting a energy and / or overview in everyday life, trying out ways to analyze and solve problems, or make gradual changes in everyday life by setting sub-goals.

Standard services in community mental health centres include appointments with psychiatrist, psychologists and/or care manager, psychoeducation, social skills training and relational support. Standard services within the rehabilitation services in Odense, Svendborg and Copenhagen include drop-in centres, self-esteems groups, peer-services, skills-training and relational support.

Data collection Baseline data is obtained by interview and questionnaires. The questionnaires are sent electronically by email or by mail. The questionnaires are returned to the researcher before randomization. In the event of failure to answer one or more items, these are reviewed by calling the participant in order to clarify any. question and get the answer complete. Healthcare services and the participants' diagnosis are obtained via the National Patient Register. Information about death is obtained from the Cause of Death Register. Meeting in MA&R will be registered by MA&R mentors, and will be returned to researcher after eight months of follow-up. At eight months of follow-up, the researcher sends questionnaires to the participants electronically or by letter, depending on what the participant prefers. Where the participants do not answer the questionnaires on their own, the participant will receive a reminder of this, by mail and / or telephone inquiry. The participant will be offered assistance from research to fill out the questionnaires. Data will be stored in REDCap. Declarations of consent will be scanned and stored on logged drives.

Fidelity Fidelity will be monitored once per course with MA&R Fidelity Scale, an instrument developed for the purpose. The evaluation will be done by external evaluators.

Sample size and power calculations

Sample size calculations is based on tracking a minimal but clinically significant difference between the intervention group and the POES-S control group (increased engagement in meaningful activities). Eklund et al. found in their RCT a small effect of 1.4 points measured on POES-S (d = 0.27) by "Balancing Everyday Life. (39) Since MA&R is of a more comprehensive format (in terms of duration and costs) than BEL, the clinically significant difference to be tracked is set to 3 points. When the standard deviation is 5.9 (39), power is 80% and the significance level is 5%, a total of 128 participants, 64 in each group must be included to track this difference.

Power calculation on the secondary outcomes is based on the fact that there are 64 participants in respectively the intervention and control group. Since it has not been possible to identify studies with the same intervention and target group as this study, the estimated effect size is based on expert opinions, systematic reviews and what is considered to be a clinically significant difference for the target group of the intervention (corresponding to a moderate effect size on d = 0.5.)

Statistics All outcome variables are continuous. The primary outcome is activity engagement, measured on POES-S. This variable will be analyzed as a continuous variable. Differences between the intervention group and the control group will be analyzed using ANOVA to determine statistical significance. Clinical significance will be calculated at Cohens d.

Multiple multivariate imputations will be used and all covariates with putative prognostic significance will be used to impute a distribution of missing data.

The continuous effect measurements will be analyzed with "repeated measurement model in mixed model analyzes with unstructured variance". The prerequisite for using this analysis and for the use of multiple imputation is that data is missing at random or data missing completely at random as opposed to non-ignorable non-response. This distinction is important because repeated measurement and multiple imputation are both models based on a statistical estimation of non-existent responses, and the preconditions for this estimation must be met in order for the assays to be valid.

We will analyze whether the conditions for using repeated measurement and multiple imputation are present by conducting a drop-out analysis. Significant prognostic characteristics of the non-followers will be compared to the participants remaining in the trial. Variables where there is a difference between participants and non-participants will be included as co-variates in the analyzes. Data analysis will be based on the intention-to-treat principle. Data from all participants will be included corresponding to the group to which they have been allocated. As a supplementary analysis, we will make per-protocol where complete cases will be analyzed.

At detailed plan for analysis will be uploaded at ClinicalTrials.gov prior analysis

ELIGIBILITY:
Inclusion Criteria:

•>18 years old

* Has disability assessment assessed by researcher at Mini-ICF Rating for Limitations of Activities and Participation in Psychological Disorders (Mini-ICF-APP) (28)
* Be diagnosed with a mental disorder and have been associated with the psychiatric treatment system, either by admission or outpatient contact.
* Has given informed consent

Exclusion Criteria:

* Diagnosed with dementia
* Have abuse as a main diagnosis, or an abuse that stands in the way of participation in MA&R
* A forensic psychiatric status
* Need for translator assistance
* Do not want to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Profiles of occupational engagement in people with severe mental illness (POES-S). | Eight months
  Activity Engagement (engagement in meaningful daily activities, social roles, and connection to the community). rating is made on nine items expressing activity engagement, for example balance between rest and activity, being able to move between places, and taking initiatives. A four-point rating schedule is used. The range is 9-36, where higher values indicate better outcome

SECONDARY OUTCOMES:
WHODAS 2.0 | Eight months
  Functioning and disability. The WHODAS 2.0, 12-item version, self-administered instrument is used. WHODAS 2.0 has two scoring options: simple and complex. Simple scoring is a hand-scoring method that does not involve weighting individual items or converting to a standardized scale.The complex scoring method is based on item-response theory and requires use of a computer program, which is available from WHO. Normative values for the WHODAS 2.0 are based on this scoring method. In WHODAS 2.0, 12 items version, Disabilities within12 domains of functioning such as social relations, household chores, participating in the community etc. are measured on a 5 point scale. 1 is no difficulties and 5 is extreme difficulties/not capable of. The scores can be summarized, to a total score reflecting level of functioning and disability. The range is 12 - 60, where lower scores indicate better outcome
Manchester Short Assessment of Quality of Life (MANSA). | Eight months
  Quality of life (MANSA) contains 16 questions. Four of them investigating objective quality of life and 12 focus on subjective quality of life, in regard to satisfaction with life as a whole, job, financial situation, friendships, leisure activities, accommodation, personal safety, people that the person lives with, family and health. Satisfaction is rated on a 7 point scale ranging from 1 which is could not be worse to 7 which is could not be better, and an overall score of subjective quality of life may be calculated. The range is 12-84, higher values indicate better outcome.
Questionnaire about Process of Recovery (QPR) | Eight months
  QPR measures aspects of the personal recovery proces, such as sense of agency and hope. The QPR has 15 items. Each item is rated on a 4-point scale (0= disagree strongly, 1=disagree, 2=neither agree nor disagree, 3=agree, 4=agree strongly). The items are summarized to a total score. The range is 0 to 70. Higher values indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, Principal Investigator — Copenhagen Research Center of Mental Health (CORE)
Locations (4):
- Denmark (4):
  - Copenhagen Socialpsychiatry, Copenhagen
  - Copenhagen Mental Health Center, Copenhagen
  - Odense kommunes rehabiliteringsteam (psychiatric rehabilitation team, Odense), Odense
  - Impuls Mødested og Kursuscenter (Drop in centre), Svendborg

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data is restricted by GDP (EU legislation)

REFERENCES:
- [Background] 1. Doroud N, Fossey E, Fortune T. Recovery as an occupational journey: A scoping review exploring the links between occupational engagement and recovery for people with enduring mental health issues. Aust Occup Ther J. 2015;62(6):378-392. 2. Gutman SA. Special issue: Effectiveness of occupational therapy services in mental health practice. Am J Occup Ther Off Publ Am Occup Ther Assoc. 2011;65(3):235. 3. Petersen KS, Bjørkedal STB, Torsting AMB, Eplov LF. Occupational Therapy Interventions in Mental Health - a scoping review of current evidence. (Submittet). 4. Eplov LF. Psykiatrisk & psykosocial rehabilitering: en recovery-orienteret tilgang. Munksgaard Danmark; 2010. 260 s. 28. Molodynski A, Linden M, Juckel G, Yeeles K, Anderson C, Vazquez-Montes M, m.fl. The reliability, validity, and applicability of an English language version of the Mini-ICF-APP. Soc Psychiatry Psychiatr Epidemiol. 2013;48(8):1347-1354. 33. Bejerholm U, Hansson L, Eklund M. Profiles of occupational engagement in people with schizophrenia (POES): the development of a new instrument based on time-use diaries. Br J Occup Ther. 2006;69(2):58-68. 34. Law H, Morrison A, Byrne R, Hodson E. Recovery from psychosis: a user informed review of self-report instruments for measuring recovery. J Ment Health. 2012;21(2):192-207. 35. Björkman T, Svensson B. Quality of life in people with severe mental illness. Reliability and validity of the Manchester Short Assessment of Quality of Life (MANSA). Nord J Psychiatry. 2005;59(4):302-306. 36. Üstün TB. Measuring health and disability: Manual for WHO disability assessment schedule WHODAS
- [Derived] Bjorkedal SB, Bejerholm U, Hjorthoj C, Moller T, Eplov LF. Meaningful Activities and Recovery (MA&R): a co-led peer occupational therapy intervention for people with psychiatric disabilities. Results from a randomized controlled trial. BMC Psychiatry. 2023 Jun 6;23(1):406. doi: 10.1186/s12888-023-04875-w. PMID 37280561
- [Derived] Bjorkedal STB, Bejerholm U, Eplov LF, Moller T. Meaningful Activities and Recovery (MA&R): the effect of a novel rehabilitation intervention among persons with psychiatric disabilities on activity engagement-study protocol for a randomized controlled trial. Trials. 2020 Sep 14;21(1):789. doi: 10.1186/s13063-020-04722-3. PMID 32928298

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03963245/SAP_000.pdf